CLINICAL TRIAL: NCT04952298
Title: EASINESS-TRIAL - An Analysis of Standardized Outcome References From an International Multicentre Cohort
Brief Title: EASINESS-TRIAL - Enhancing Safety in Epilepsy Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Erlangen-Nürnberg (Other); University Clinic Frankfurt (Other); Vienna General Hospital (Other)
Responsible Party: Principal Investigator, Richard Drexler, Resident, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: EASINESS
Record Dates: First submitted 2021-06-11; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy, Temporal Lobe; Amygdalo-Hippocampal Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mesial temporal lobe epilepsy surgery — Medial temporal lobe epilepsy surgery including
  * selective Amygdalohippocempectomy (SAH) including anterior parahippocampal gyrus / entorhinal cortex
  * anteromedial temporal lobe resection including amygdalohippocampectomy
  * anterior temporal lobe resection

SUMMARY:
To conduct a retrospective multicenter cohort study to define surgical benchmark values for best achievable outcomes following surgery for mesial temporal lobe epilepsy. Established benchmark serve as reference values for the evaluation of future surgical strategies and approaches.

DETAILED DESCRIPTION:
Surgeons strive for the best possible outcome of their surgeries with the greatest possible chance for recovery of the patients. Therefore, monitoring and quality improvement is increasingly important in surgery. For this purpose, different concepts were developed with the aim to assess best achievable results for several surgical procedures and reduce unwarranted variation between different centers. The most common used concept in surgery is a combination of various clinical indicators with a focus on treatment and adverse events which offers a more reliable analysis than single-outcome indicators. The concept of a benchmark establishes reference values which represents the best possible outcome of high-volume centers and can be used for comparison and improvement. Benchmark values are established within a patients' cohort for which the best possible outcome can be expected. The aim of our study is the establishment of robust and standardized outcome references after amygdalohippocampectomy for temporal lobe epilepsy. After successful implantation of benchmarks from an international cohort of renowned centers, these data serve as reference values for the evaluation of novel surgical techniques and comparisons among centers or future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Centres with ≥30 seizure-specific resections (excluding vagus nerve stimulation) as an average per year during the 5-year study period
* Patients who went through mesial temporal lobe epilepsy surgery

Exclusion Criteria:

* Only neocortical temporal resection
* Recurrent resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who went through medial temporal lobe epilepsy surgery at high-volume centres
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Seizure Outcome | up to 1 year
  International League Against Epilepsy (ILAE) Outcome Scale
  - Class 1 (seizure-free) to class 6 (>100% increase of baseline seizure days)
Figural memory | up to 1 year
  Improvement, unchanged, deterioration, e.g. at the Rey Auditory-Verbal Learning Test
Attention | up to 1-year
  Improvement, unchanged, deterioration, e.g. at the Wechsler Memory Scale
Verbal memory | up to 1 year
  Improvement, unchanged, deterioration, e.g. at the Rey Auditory-Verbal Learning Test
Neurological deficit | up to 1 year
  None, visual field loss, diplopia, motor deficit, sensory deficit, language impairment (according to NANO scale)
3D-Volumetry of extent of resection on MRI | 3 months postoperatively
Number of anticonvulsive drugs | up to 1 year
Reoperation | up to 1 year
Temporalis muscle atrophy | up to 1 year
  Not-visible or visible
Complication of any severity | up to 1 year
Stroke | up to 1 year
Surgical site infection | up to 1 year
In-hospital mortality after index surgery | up to 1 year
Length of ICU stay after index surgery | up to 1 year
Length of stay after index surgery | up to 1 year

OTHER OUTCOMES:
Age | At time of surgery
Sex | At time of surgery
Education status | At time of surgery
American Society of Anaesthesiologists (ASA) physical status | At time of surgery
  1 (healthy person) to 6 (declared brain-dead person)
Body mass index | At time of surgery
  in kg/m^2
History of neonatal seizures | At time of surgery
History of febrile seizures | At time of surgery
History of encephalitis or meningitis | At time of surgery
Congestive heart failure | At time of surgery
Coagulopathy / bleeding disorder | At time of surgery
Diabetes mellitus | At time of surgery
Age at epilepsy onset | At time of surgery
Type of seizures | At time of surgery
Average monthly frequency of seizures impairing awareness in year before surgery | At time of surgery
Number of anticonvulsive drugs | At time of surgery
Neurological deficit | At time of surgery
  None, visual field loss, diplopia, motor deficit, sensory deficit, language impairment (according to NANO scale)
Preoperative MRI lesion | At time of surgery
MRI post-processing conducted | At time of surgery
Additional preoperative diagnostic tool | At time of surgery
  PET, SPECT, MEG, Wada test
Type of surgery | Surgery
  Selective amygdalohippocampectomy, anteromedial temporal lobe resection including amydalohippocampectomy, anterior temporal lobe resection
Intraoperative navigation | Surgery
  No or yes
Side of procedure | Surgery
Operating duration | Surgery
  minutes
Histological finding | At time of surgery
  Hippocampal sclerosis, focal cortical dysplasia, dysembryoplastic neuroepithelial tumours, Ganglioglioma, others

CONTACTS AND LOCATIONS:
Overall Officials: Richard Drexler, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided